CLINICAL TRIAL: NCT05624736
Title: Artificial Intelligence Research of Hierarchical Diagnosis for Adult Diffuse Glioma Based on Deep Learning
Brief Title: Hierarchical Diagnosis for Adult Diffuse Glioma Based on Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-MS-25
Record Dates: First submitted 2022-11-13; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-07

CONDITIONS: Astrocytoma; Glioblastoma Multiforme; Oligodendroglioma
Keywords: Astrocytoma; Glioblastoma; Oligodendroglioma; deep learning; artificial intelligence
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Oligodendroglioma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Glioblastoma Group: Patients with the diagnosis of Glioblastoma based on 2021 WHO central nervous system tumor guideline.
  Interventions: Diagnostic Test: multi-parametric magnetic resonance imaging scan; Diagnostic Test: Pathology examination
- Astrocytoma Group: Patients with the diagnosis of Astrocytoma based on 2021 WHO central nervous system tumor guideline.
  Interventions: Diagnostic Test: multi-parametric magnetic resonance imaging scan; Diagnostic Test: Pathology examination
- Oligodendroglioma Group: Patients with the diagnosis of Oligodengroglioma based on 2021 WHO central nervous system tumor guideline.
  Interventions: Diagnostic Test: multi-parametric magnetic resonance imaging scan; Diagnostic Test: Pathology examination

INTERVENTIONS:
Diagnostic Test: multi-parametric magnetic resonance imaging scan — Pre-operative multi-parametric magnetic resonance imaging scans including T1WI, T2WI, T1CE, FLAIR and DWI were taken for clinical needs.
Diagnostic Test: Pathology examination — The tumor specimen obtained from the surgery were sent to the pathology department for histopathologic examination, immunohistochemistry and gene sequencing test

SUMMARY:
This is a restrospective study to establish a deep learning model based on multi-parametric magnetic resonance imaging scans to predict Grade, histopathologic type and genotype of adult diffuse Glioma.

DETAILED DESCRIPTION:
Glioma is a common kind of tumor in central nervous system. The pre-operative prediction of grade, histopathologic type and genotype is important for treatment and management of Adult diffuse Glioma patients. Right now, most of the diagnostic prediction models on glioma are based on 2016 WHO central nervous system tumor guideline. The goal of this study is to establish a new deep learning model to predict Grade, histopathologic type and genotype of adult diffuse Glioma. We will recruit 500 patients with pathologically confirmed diagnosis of Glioblastoma, Astrocytoma and Oligodendroglioma who received neurologic surgery in our center. Each subject underwent pre-operative multi-parametric magnetic resonance imaging scans including T1WI, T2WI, T1CE, FLAIR and DWI. Pathologic diagnosis of each patient are available in pathology department. A deep learning based hierarchical diagnosis

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery in Nanjing DrumTower Hospital between 2010.01 and 2022.05 with post-surgery pathological diagnosis of WHO Grade II to IV Adult Diffuse Glioma.
2. Available pre-surgery T1WI, T2WI, T1CE, FLARI and DWI MR sequences
3. No pre-surgery anti-tumor therapy

Exclusion Criteria:

1. Poor image quality
2. Failed image preprocessing
3. Unavailable pathology data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of adult diffuse glioma who recevived tumor rection surgery in our center
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Grade | up to 2 weeks
  Tumor Grade based on 2021 WHO central nervous system tumor guideline
Tumor Histologic diagnosis | up to 2 weeks
  Tumor histologic diagnosis based on 2021 WHO central nervous system tumor guideline
Tumor genotype | up to 2 weeks
  Tumor genotype based on 2021 WHO central nervous system tumor guideline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
We don't plan to share IPD with other researches